CLINICAL TRIAL: NCT01088607
Title: Ursodeoxycholic Acid Therapy in Pediatric Primary Sclerosing Cholangitis: A Pilot Withdrawal/Reinstitution Trial
Brief Title: Safety and Efficacy Study of Ursodeoxycholic Acid Therapy in Pediatric Primary Sclerosing Cholangitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); University of Colorado, Denver (Other); University of California, San Francisco (Other); University of Pittsburgh (Other); Phoenix Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Children's Healthcare of Atlanta (Other); Children's Hospital Los Angeles (Other); Baylor College of Medicine (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD-003709
Record Dates: First submitted 2010-03-12; First posted 2010-03-17 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Primary sclerosing cholangitis; Autoimmune hepatitis; Cholestatic liver disease; Cirrhosis; Children; Primary Sclerosing Cholangitis/Autoimmune Hepatitis Overlap
MeSH Terms: conditions — Cholangitis, Sclerosing; Hepatitis, Autoimmune; Fibrosis | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UDCA Withdrawal and Reinstitution (Experimental): Each study subject will undergo serial UDCA withdrawal and reinstitution.
  Interventions: Drug: ursodeoxycholic acid (UDCA)

INTERVENTIONS:
Drug: ursodeoxycholic acid (UDCA) — Pediatric PSC patients already receiving UDCA therapy will enter a four-phase trial consisting of baseline data collection (phase I, 4 weeks), 50% reduction in UDCA dose (phase II, 4 weeks), discontinuation of UDCA (phase III, 8 weeks) and reinstitution of therapy at a dose of 20 mg/kg/day (phase IV, 8 weeks). Surveillance and endpoint evaluation for each phase will include liver chemistries and clinical data. Comparisons will be made between baseline and the end of phase III (primary outcome) and between the end of phase III and the end of phase IV (secondary outcome). Serum cytokine biomarkers will be measured and compared between baseline and the end of phase III and between the end of phases III and IV.
  Other Names: Ursodeoxycholic acid; URSO 250; URSO Forte; Actigall; Ursodiol; UDCA

SUMMARY:
Primary sclerosing cholangitis (PSC), although uncommon, is a devastating and insidiously progressive liver disease, resulting from advancing inflammation, fibrosis and obliteration of the bile ducts in the liver, leading to cirrhosis and end-stage liver disease. Although prognosis in children may be somewhat better than that of adults, approximately one third of pediatric patients require transplantation by adulthood. Other than transplantation, there is to date no therapy conclusively proven to improve the long-term outcome. Ursodeoxycholic acid (UDCA) improves biochemical markers of liver disease, although in high doses does not clearly improve the long-term outcome in adults, and in a recent study may have actually worsened outcome. Childhood PSC is different from that of adult PSC in many ways, and children may derive more short-term, as well as long-term, benefit than adults. This unique multicenter study will carefully monitor the effects of withdrawal and restarting UDCA on liver injury and inflammation in children with PSC. The preliminary data will help in the design of a more definitive larger study to determine if UDCA has a beneficial role in the treatment of PSC in children. Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Primary sclerosing cholangitis (PSC), a devastating and insidiously progressive cholestatic liver disease, results from advancing inflammation, fibrosis and obliteration of the intra- and extrahepatic bile ducts, leading to cirrhosis and end-stage liver disease. PSC is an uncommon disorder (prevalence in the US of 8-14/100,000 with even lower prevalence in children). Although prognosis in children may be somewhat better, approximately one third of pediatric patients require transplantation by adulthood. Other than transplantation, there is to date no therapy conclusively proven to improve the long-term outcome. Ursodeoxycholic acid (UDCA) improves biochemical markers of liver disease, although in high doses does not clearly improve the long-term outcome in adults. Furthermore, a recent large adult trial of high-dose UDCA therapy suggested a higher incidence of serious adverse events and poor outcomes with UDCA treatment, leading many centers to discontinue UDCA therapy in adult patients. Childhood PSC is different from the adult disease including a stronger association with both autoimmune markers and histologic features and a trend to higher transaminases at diagnosis. Furthermore, in response to intermediate-dose UDCA therapy, there is a more striking and prompt improvement in biochemistries as compared to adults. In light of the prompt normalization of liver enzymes and the fact that UDCA is well tolerated in children, pediatric hepatologists are reluctant to generalize the adult UDCA study results to children and to stop UDCA therapy. This presents a significant dilemma: Should UDCA therapy be stopped in pediatric PSC patients to avoid a possible adverse influence on long-term prognosis at the risk of losing a possible beneficial effect on disease progression in children? Additional factors in children with PSC/autoimmune hepatitis (AIH) overlap are the long-term adverse effects of corticosteroids and azathioprine use. If UDCA therapy is effective as monotherapy, these complications may be avoided. Therefore, we propose a preliminary UDCA withdrawal and reinstitution trial in pediatric PSC patients to collect data to support the design of a larger, longer-term randomized, placebo-controlled trial of UDCA therapy in childhood PSC. This pilot study, which will utilize the infrastructure and participating centers of the STOPSC (Studies of Primary Sclerosing Cholangitis) consortium, will test the following hypotheses: 1) UDCA therapy yields a rapid biochemical response in children with PSC, thus withdrawal would lead to increased biochemical evidence of disease. 2) UDCA therapy suppresses liver and biliary inflammation in children with PSC, thus withdrawal of therapy would result in a burst of inflammatory activity and an increase in serum cytokine biomarkers, 3) Biochemical control of childhood PSC with histologic features of AIH is dependent upon treatment with immunosuppression in addition to UDCA, therefore childhood PSC without histologic features of AIH will worsen significantly with UDCA withdrawal compared to PSC with histological features of AIH.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female < 21 years of age, no racial or ethnic restrictions
2. Pediatric PSC diagnosed as per the criteria developed by STOPSC (2 of 3 required):

   * Serum GGT increased more than 50% above the upper limit of normal for age
   * Endoscopic retrograde cholangiopancreatography (ERCP), percutaneous transhepatic cholangiography (PTC) or magnetic resonance cholangiopancreatography (MRCP) findings of intrahepatic and/or extrahepatic bile duct irregularities consistent with PSC
   * Liver biopsy abnormalities consistent with chronic biliary injury Note that these criteria will include patients with small duct PSC who have normal biliary imaging with the required biochemical and histologic criteria.
3. Patients with PSC/AIH overlap will also be included who meet the criteria for PSC plus have liver histologic features of AIH.
4. Biochemically quiescent liver disease defined by an ALT and GGT < 2.0 X upper limit of normal (ULN) measured on two separate occasions > 2 weeks apart
5. Prior and on-going UDCA therapy at a dose of at least 13 mg/kg/day or 600 mg/day for more than 6 months
6. Ability to swallow pills
7. Quiescent inflammatory bowel disease (IBD) as reflected by a modified Pediatric Ulcerative Colitis Activity Index score of less than 6 or a modified Pediatric Crohn's Disease Activity Index score of less than 15.
8. Not excluded by the STOPSC pediatric PSC exclusion criteria (see Appendix) that are designed to minimize misdiagnosis due to other primary liver diseases, previous biliary injury/surgery, therapies, or systemic disorders that may secondarily affect the liver and/or biliary tract.
9. Subjects will remain on all current medications, including those for IBD and immunosuppressive therapy.
10. Female subjects of childbearing age will be required to have a pregnancy test, and if sexually active, will be required to use an accepted method of birth control during the course of the study.
11. Parent or legal guardian must be willing to provide signed and dated informed consent documentation. Assent from the child or adolescent will be obtained as appropriate.

Exclusion Criteria:

1. Evidence of decompensated cirrhosis:

   * Cirrhosis as defined by biopsy findings or evidence of portal hypertension with no other known cause and:

     * Platelet count < 100,000 or,
     * Spleen palpable more than 2 cm below the left costal margin or,
     * Ascites or,
     * Varices or other GI manifestation of portal hypertension
   * Decompensated liver disease defined by:

     * Serum total bilirubin (TB) > 5 mg/dl and direct bilirubin (DB) > 1 mg/dl or,
     * Prothrombin time (PT) prolonged by more than 3 seconds after parenteral vitamin K administration or,
     * Ascites requiring diuretic therapy or,
     * Serum albumin < 3 g/dl
2. Evidence of acute liver failure:

   * No prior history of liver disease and
   * PT > 20 seconds or INR > 2.0 unresponsive to parenteral vitamin K administration or,
   * PT > 15 seconds or international normalized ratio (INR) > 1.5 with change in mental status ascribable to hepatic encephalopathy
3. History of cholangitis or bile duct strictures requiring intervention
4. Liver transplantation

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the change in alanine aminotransferase (ALT), gamma-glutamyl transpeptidase (GGT) or biomarkers for inflammation in study subjects at baseline compared to the end of Phase III (UDCA discontinuation) of the study. | 16 weeks
  Phase I-4 weeks, Phase II-4 weeks, Phase III-8 weeks, Phase IV-8 weeks

SECONDARY OUTCOMES:
A secondary outcome will be the change in ALT, GGT or biomarkers for inflammation in study subjects at the end of Phase III (UDCA discontinuation) compared to the end of Phase IV (UDCA reinstitution) of the study. | 8 weeks
  Phase I-4 weeks, Phase II-4 weeks, Phase III-8 weeks, Phase IV-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis D Black, M.D., Principal Investigator — University of Tennessee; Benjamin Shneider, M.D., Principal Investigator — Baylor College of Medicine
Locations (12):
- United States (12):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Children's Healthcare of Atlanta, Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas